CLINICAL TRIAL: NCT00889733
Title: A Phase I/II Trial of Intraperitoneal (IP) Cisplatin Combined With IV Paclitaxel in Patients With Epithelial Ovarian Cancer Optimally Debulked at Their Initial Surgery Performed Following Neoadjuvant Intravenous Chemotherapy
Brief Title: Intraperitoneal (IP) Cisplatin Given With Paclitaxel to Treat Epithelial Ovarian Cancer
Acronym: OVHM-01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OVHM-01
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Infusions, Parenteral; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IP Cisplatin (Experimental): Patients with epithelial ovarian cancer who have undergone optimal debulking surgery receive IP Cisplatin with IV Paclitaxel.
  Interventions: Drug: Intraperitoneal (IP) Cisplatin

INTERVENTIONS:
Drug: Intraperitoneal (IP) Cisplatin — For patients who have had neoadjuvant chemotherapy followed by optimal debulking surgery they go on to receive combined IP Cisplatin and IV Paclitaxel.

SUMMARY:
The purpose of this study is to determine whether intraperitoneal (IP) Cisplatin combined with intravenous (IV) Paclitaxel is well tolerated in women with epithelial ovarian cancer who have had neoadjuvant chemotherapy followed by initial debulking surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven epithelial ovarian cancer
* Previously received no more than 4 cycles of neoadjuvant platinum based chemotherapy, followed by debulking surgery
* ECOG PFS <_ 2
* Adequate haematological (absolute neutrophil count >_ 1,500/mm3; platelets >_ 100,000/mm3; hemoglobin >_ 100g/L); renal (<_ upper limit of normal) and hepatic function
* Age >_ 18 years
* Written informed consent and the ability of the patient to co-operate with treatment and follow up

Exclusion Criteria:

* Contraindication to platinum/Paclitaxel chemotherapy: prior anaphylaxis to Carboplatin/Paclitaxel, unresolved or excessive toxicity from neoadjuvant chemotherapy. Patients must not have suffered significant bone marrow suppression during prior treatment. The significance of previous treatment delay and/or dose modification is to be determined by the Principle Investigator on a patient-by-patient basis.
* Serious concomitant medical condition, which in the investigators opinion would not make the patient a good candidate for the clinical trial.
* Patients with a past or concomitant malignancy other than skin cancer (excluding melanoma)
* Patients known to be serologically positive for Hepatitis B, C or HIV
* History of congestive heart failure or unstable angina or those who had a myocardial infarction within the past 6 months. Patients who were not expected to tolerate the hemodynamic effects of the fluid administered as part of the IP protocol.
* Patients who have not received chemotherapy prior to surgery
* Greater than 6 weeks from time of surgery to commencement of IP chemotherapy
* Residual disease greater than 1 cm at time of surgery. Patients whom in the surgeon's opinion are candidates for such surgery may be consented preoperatively to allow intraoperative IP catheter insertion. If however the surgeon is not able to reduce the bulk of disease to less than or equal to 1 cm, patients will be removed from the study and an IP catheter SHOULD NOT be placed.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and Dose Tolerance | Day 1 of each cycle and assessed every 3 months in follow-up (if applicable)

SECONDARY OUTCOMES:
Time to progression | Day 1 of cycle 1 & 2 and every 3 months in follow-up until progression noted

CONTACTS AND LOCATIONS:
Overall Officials: Helen MacKay, MD, Principal Investigator — UHN - Princess Margaret Cancer Centre
Locations (1):
- University Health Network - Princess Margaret Hospital, Toronto, Ontario, Canada